CLINICAL TRIAL: NCT01353339
Title: Quinolone Prophylaxis for the Prevention of BK Virus Infection in Kidney Transplantation: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); St. Paul's Hospital, Canada (Other); Vancouver General Hospital (Other); University of Alberta (Other); University of Manitoba (Other); University Health Network, Toronto (Other); Unity Health Toronto (Other); St. Joseph's Healthcare Hamilton (Other); London Health Sciences Centre (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIHR MOP 222493, 2010-292
Record Dates: First submitted 2011-05-11; First posted 2011-05-13 (Estimated); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2014-10

CONDITIONS: Disease Due to BK Polyomavirus; Kidney Transplant Infection
Keywords: Kidney Transplant; BK Polyomavirus Infection
MeSH Terms: interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sugar pill (Placebo Comparator)
  Interventions: Drug: Levofloxacin
- levofloxacin (Active Comparator)
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin — 500mg, PO, once daily for 3 months
  Other Names: Apo-levofloxacin; DIN 02284707

SUMMARY:
Primary Research Questions:

Efficacy, safety and feasibility of a 3-month course of levofloxacin in a pilot study will be assessed.

1. Under efficacy, this pilot will determine whether levofloxacin can decrease the incidence of BK viruria and peak urine BK viral load.
2. Under safety, this pilot will determine the incidence of adverse events with levofloxacin.
3. Under feasibility, this pilot will determine the number of kidney transplant patients randomized over an eight month enrolment period, adherence to the levofloxacin and frequency of patient drop-out and loss to follow-up

DETAILED DESCRIPTION:
BK virus infection has emerged as a major complication in renal transplantation leading to a significant reduction in graft survival. There are currently no proven strategies to prevent or treat BK virus infection. Quinolone antibiotics, such as levofloxacin, have demonstrated activity against BK virus. The investigators hypothesize that administration of a quinolone antibiotic, when given early post-transplantation, will prevent the establishment of BK viral replication in the urine and thus prevent systemic BK virus infection. A non-randomized study in kidney transplant recipients found that patients given levofloxacin or ciprofloxacin had a significantly lower incidence of BK viremia compared to those not receiving a quinolone (4% versus 24.5%, P=0.02).

Objective: The primary objective of the full trial will be to determine if the quinolone levofloxacin decreases the occurrence of doubling creatinine, transplant failure or death in kidney transplant recipients. The aim of this pilot trial is to assess the efficacy, safety and feasibility of a 3-month course of levofloxacin in the kidney transplant population.

Results from this pilot study will provide vital information to design and conduct a large, multi-centre trial to determine if quinolone therapy decreases meaningful clinical outcomes in kidney transplantation. If levofloxacin significantly reduces BK viruria and urine viral loads in kidney transplantation it will provide important justification of biologic effect to progress to the larger trial. If the full trial shows that levofloxacin significantly reduces BK infection and improves outcomes, its use in renal transplantation will be strongly endorsed given the lack of proven therapies for this condition.

ELIGIBILITY:
Inclusion Criteria:

* a primary or repeat kidney transplant recipient (deceased or living donor)
* age greater or equal to 18 years

Exclusion Criteria:

* Unable to provide informed consent
* Greater than 5 days post-transplantation
* BK virus nephropathy with a previous transplant
* History of allergic reaction to any quinolone antibiotic
* History of quinolone associated tendonitis or tendon rupture
* Corrected QT interval prolongation on EKG as defined by Al-Khatib
* Concomitant use of medication known to prolong the QT interval such as class IA antiarrhythmic drugs (e.g. quinidine, procainamide, disopyramide), class III antiarrhythmic drugs (e.g. amiodarone, sotalol), azole antifungals (e.g. fluconazole) or macrolide antibiotics (e.g. erythromycin)
* Pregnant or breastfeeding as safety of levofloxacin not established
* Requires quinolone antibiotic for more than 14 days (e.g. for UTI prophylaxis)
* Recipient of a multi-organ transplant (e.g. kidney-pancreas)
* Currently enrolled in another interventional trial
* Previously enrolled in this study
* History of rhabdomyolysis
* Significant allergic reaction to ≥ 3 classes of antibiotics as these patients may have no other option other than quinolones for routine infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2014-02-25 (Actual); Study Completion 2014-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Knoll, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (11):
- Canada (11):
  - Capital Health - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Winnipeg Health Science Center, Winnipeg, Manitoba
  - QEII Health Science Center, Halifax, Nova Scotia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - London Health Science Center, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec

REFERENCES:
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091
- [Derived] Knoll GA, Humar A, Fergusson D, Johnston O, House AA, Kim SJ, Ramsay T, Chasse M, Pang X, Zaltzman J, Cockfield S, Cantarovich M, Karpinski M, Lebel L, Gill JS. Levofloxacin for BK virus prophylaxis following kidney transplantation: a randomized clinical trial. JAMA. 2014 Nov 26;312(20):2106-14. doi: 10.1001/jama.2014.14721. PMID 25399012
- [Derived] Humar A, Gill J, Johnston O, Fergusson D, House AA, Lebel L, Cockfield S, Kim SJ, Zaltzman J, Cantarovich M, Karpinski M, Ramsay T, Knoll GA. Quinolone prophylaxis for the prevention of BK virus infection in kidney transplantation: study protocol for a randomized controlled trial. Trials. 2013 Jun 21;14:185. doi: 10.1186/1745-6215-14-185. PMID 23800312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was randomized on December 1, 2011, and recruitment continued until June 25, 2013. The last patient follow-up visit was February 25, 2014.
Pre-assignment Details: Eligible patients with written informed consent were randomly assigned to receive either levofloxacin or placebo in a 1:1 fashion. Allocation was achieved through web-based central randomization in variable blocks stratified by center. An independent statistician prepared the randomization schemes. Physicians, nurses, investigators, and research staff were blinded to the randomization scheme, and active study medication and matching placebo were identical in appearance
Period: Overall Study
Arm/Group | Levofloxacin | Sugar Pill
Started | 76 | 78
Discontinued Intervention | 12 | 14
Incomplete Follow-up | 22 | 28
Completed | 76 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants were randomized in the study and included in baseline analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin | Sugar Pill | Total
Number analyzed (Participants) | 76 | 78 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (14.2) | 48.2 (12.7) | 48 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 16 | 43
  Male | 49 | 62 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 49 | 50 | 99
  Black | 3 | 7 | 10
  Asian | 3 | 7 | 10
  Aboriginal | 4 | 1 | 5
  Other | 14 | 11 | 25
  Unknown | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 76 | 78 | 154

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of BK Viruria
Description: BK viruria was defined as 500 copies/mL or more of BK virus DNA in the urine.
Time Frame: 12 months post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 22 | 26

2. Secondary Outcome: Adverse Events
Description: Incidence and type of all adverse events
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 27 | 29

3. Secondary Outcome: Acute Rejection
Description: Incidence of Acute rejection
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 6 | 5

4. Secondary Outcome: Clostridium Difficile Associated Diarrhea
Description: Incidence of microbiologically confirmed clostridium difficile associated diarrhea
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 36 | 30

5. Secondary Outcome: Infections
Description: Incidence of other infections (viral, bacterial and fungal) based on established guidelines
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of infections per patient
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Number of infections per patient | 1.4 (1.6) | 1.3 (2.2)

6. Secondary Outcome: Quinolone Resistance
Description: Incidence of quinolone resistance where a quinolone would have been a therapeutic option
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 14 | 15

7. Secondary Outcome: Allograft Loss
Description: Absence of kidney function in allograft
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 0 | 1

8. Secondary Outcome: Mortality
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 0 | 0

9. Secondary Outcome: Adherence
Description: Proportion of randomized participants who are adherent to the protocol.
Time Frame: 12 months
Measure: Number; unit: Percentage of participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Percentage of participants | 68.5 | 70.4

10. Secondary Outcome: Use of Quinolones
Description: Use of quinolones outside of the protocol
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 19 | 14

11. Secondary Outcome: Proportion of Patient Drop-out and Loss to Follow-up
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 0 | 0

12. Secondary Outcome: Quantitative BK Urine Viral Load
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
copies/mL | 7550 (16542) | 4503 (5419)

13. Secondary Outcome: BK Viremia
Description: BK viremia defined as ≥250 copies/mL of BK virus DNA in the plasma
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin | Sugar Pill
Number analyzed (Participants) | 76 | 78
Participants | 6 | 9

ADVERSE EVENTS:
Arm/Group | Levofloxacin | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/78
Serious Adverse Events (participants affected / at risk) | 6/76 | 1/78
Other Adverse Events (participants affected / at risk) | 76/76 | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levofloxacin (N=76) | Sugar Pill (N=78)
tendinitis (Musculoskeletal and connective tissue disorders) | 6 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levofloxacin (N=76) | Sugar Pill (N=78)
Hospitalization (General disorders) | 22 | 26
Over 1 infection (Infections and infestations) | 45 | 35
Culture-positive infections (Infections and infestations) | 30 | 46
Diarrhea (Gastrointestinal disorders) | 36 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No